CLINICAL TRIAL: NCT05805293
Title: High-Velocity Nasal Insufflation Therapy Versus Non-Invasive Ventilation In Management Of Acute Hypercapnic Respiratory Failure In Obesity Hypoventilation Syndrome: A Randomized Controlled Trial
Brief Title: HVNI Versus NIV In Management Of Acute Hypercapnic Respiratory Failure In OHS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rofaida Raafat Talaat Ibrahim, Assistant lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HVNI versus NIV in OHS
Record Dates: First submitted 2023-03-25; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Obesity Hypoventilation Syndrome (OHS)
MeSH Terms: conditions — Obesity Hypoventilation Syndrome | interventions — Noninvasive Ventilation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-Velocity Nasal Insufflation (Experimental)
  Interventions: Device: High-Velocity Nasal Insufflation Therapy
- Non-Invasive ventilation (Experimental)
  Interventions: Device: Non-Invasive Ventilation

INTERVENTIONS:
Device: High-Velocity Nasal Insufflation Therapy — Parameter settings for the HVNI apparatus are as follows:
  1. The flow of HVNI will initially be set at 30-40 L/min, and inspiratory flow rate could be increased to 45-60 L/min.
  2. FIO2 will be adjusted to maintain a SaO2 more than 90 % and relative humidity of 30-34%.
  3. Temperature range of 35-37°C.
  Arms: High-Velocity Nasal Insufflation
Device: Non-Invasive Ventilation — Patients will be put on inspiratory/expiratory pressure 10/5 cmH2O (11). The inspiratory and expiratory pressures will be titrated with increments of 2 cmH2O based on improvement of oxygen saturation by continuous pulse oximetry and arterial blood gases values, alleviation of dyspnea and a decrease of respiratory rate and heart rate. The maximum allowed inspiratory pressure was 20 cm H2O. The maximum allowed expiratory pressure was 10 cm H2O.
  Arms: Non-Invasive ventilation

SUMMARY:
1. Assessment of benefits of HVNI in management of obesity hypoventilation syndrome complicated with acute hypercapnic respiratory failure.
2. Compare the value, safety and effectiveness of HVNI and NIV in patients with obesity hypoventilation syndrome complicated with acute hypercapnic respiratory failure.

DETAILED DESCRIPTION:
Obesity has become a worldwide health concern. Moreover, obese patients often present comorbidities, such as obstructive apnea syndrome or obesity hypoventilation syndrome. Atelectasis formation is increased in obese patients, because of the negative effects of thoracic wall weight and abdominal fat mass on pulmonary compliance, leading to decreased functional residual capacity (FRC) and arterial oxygenation. The repetitive occurrence of rapid eye movement (REM) sleep, hypoventilation or obstructive sleep apnea with long-lasting apnea and hypopnea induces a secondary depression of respiratory drive with daytime hypercapnia, leading to obesity hypoventilation syndrome. Obesity hypoventilation syndrome is defined as a combination of obesity (body mass index [BMI] ≥ 30 kg/m2), daytime hypercapnia (PaCO2 > 45 mm Hg), and disordered breathing during sleep.

Obese patients represent a specific population in the intensive care unit. Obese patients can be admitted in a critical care setting for de novo acute respiratory failure, 'acute-on-chronic' respiratory failure with an underlying disease, such as an obesity hypoventilation syndrome, or in the perioperative period. The main challenges for ICU clinicians are to take into account the pulmonary pathophysiological specificities of the obese patient to optimize airway management and non-invasive or invasive mechanical ventilation.

Noninvasive ventilation (NIV) has revolutionized the management of acute respiratory failure. NIV obviates endotracheal intubation and thus decreases the risk of ventilator-induced pneumonia, shortens ICU stay, and decreases the overall cost of hospitalization.

Oxygen delivery through high flow nasal cannula (HFNC) has used for the treatment of certain hypoxic situations like bronchiolitis in neonate. HFNC acts as non-invasive ventilator by reducing airway resistance and improving CO2 clearance by providing positive end-expiratory pressure (PEEP). Therefore, it is feasible to employ NFC in the case of obstructive pulmonary diseases. Since HFNC can open the airway by inducing stenting effects, it supplies more effective oxygenation with stable fraction of inspired oxygen (FIO2) in the range of 21 to 100% and a flow rate of up to 60 L/min.

High velocity nasal insufflation (HVNI), a form of HFNC that utilizes a small-bore nasal cannula to generate higher velocities of gas delivery than its counterparts using large bore HFNC, has the ability to accomplish complete purge of extra thoracic dead space at flow rates of 35 liters/min and may be able to provide ventilatory support in patients with acute hypercapnic respiratory failure in addition to oxygenation support.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years.
2. Obesity hypoventilation syndrome with acute hypercapnic respiratory failure. A) Body mass index [BMI] ≥ 30 kg/m2. B) Daytime hypercapnia (PaCO2 > 45 mm Hg) C) PH < 7.35 D) Arterial oxygen saturation (SaO2) <90%

Exclusion Criteria:

1. Age <18 years.
2. Pulmonary infiltrates suggesting pulmonary edema, pneumonia, active tuberculosis, or its sequelae.
3. Patients with gas exchange alterations due to other conditions, such as bronchiectasis, fibrosis of the pleural space (fibrothorax), neuromuscular disease and chronic obstructive pulmonary disease (COPD)
4. Pregnancy.
5. Contraindications for positive-airway pressure devices.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Improvement of hypercapnia and oxygenation | Baseline
  decrease rate of invasive mechanical ventilation and mortality

REFERENCES:
- [Background] Masa JF, Pepin JL, Borel JC, Mokhlesi B, Murphy PB, Sanchez-Quiroga MA. Obesity hypoventilation syndrome. Eur Respir Rev. 2019 Mar 14;28(151):180097. doi: 10.1183/16000617.0097-2018. Print 2019 Mar 31. PMID 30872398
- [Background] Chawla R, Dixit SB, Zirpe KG, Chaudhry D, Khilnani GC, Mehta Y, Khatib KI, Jagiasi BG, Chanchalani G, Mishra RC, Samavedam S, Govil D, Gupta S, Prayag S, Ramasubban S, Dobariya J, Marwah V, Sehgal I, Jog SA, Kulkarni AP. ISCCM Guidelines for the Use of Non-invasive Ventilation in Acute Respiratory Failure in Adult ICUs. Indian J Crit Care Med. 2020 Jan;24(Suppl 1):S61-S81. doi: 10.5005/jp-journals-10071-G23186. PMID 32205957
- [Background] Fernandez Alvarez R, Belda Ramirez J, Rubinos Cuadrado G, Buchelli Ramirez H, Fole Vazquez D, Iscar Urrutia M, Rodriguez Jerez F, Vazquez Lopez MJ, Casan Clara P. Obesity-Hypoventilation Syndrome: Baseline Hemodynamic Status and Impact of non-Invasive Ventilation. Arch Bronconeumol (Engl Ed). 2020 Jul;56(7):441-445. doi: 10.1016/j.arbres.2019.08.022. Epub 2019 Dec 25. English, Spanish. PMID 31882192
- [Background] Nicolini A, Ferrando M, Solidoro P, Di Marco F, Facchini F, Braido F. Non-invasive ventilation in acute respiratory failure of patients with obesity hypoventilation syndrome. Minerva Med. 2018 Dec;109(6 Suppl 1):1-5. doi: 10.23736/S0026-4806.18.05921-9. PMID 30642143